CLINICAL TRIAL: NCT04379505
Title: Palliative Expeditiously Adaptive Quad Shot Radiation Therapy (PEAQ-RT): A Pilot Study of Consolidated Simulation and Target Identification of Quad Shot Radiation Therapy Using an Adaptive Radiotherapy Workflow With a Novel Ring Gantry Radiotherapy Device
Brief Title: Palliative Expeditiously Adaptive Quad Shot Radiation Therapy (PEAQ-RT)
Acronym: PEAQ-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 202004210
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Particle Accelerators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Quad shot radiation (Experimental): -Radiotherapy will consist of Quad shot radiation delivered on the Ethos ring gantry kV-CBCT combined with linear accelerator system to a dose of 14 Gy in four, twice-daily fractions of 3.5 Gy delivered at least 6 hours apart over two days for a possible total of 3 cycles delivered in 3 to 4 intervals for a cumulative dose of of 42 Gy in 12 fractions. Cycle 2 and 3 of treatment is not mandated per protocol but may be given at the discretion of the treating physician.
  Interventions: Device: Ring gantry kV-CBCT combined with linear accelerator (Halcyon); Radiation: Quad shot radiation

INTERVENTIONS:
Device: Ring gantry kV-CBCT combined with linear accelerator (Halcyon) — -Varian Medical Systems is the manufacturer
Radiation: Quad shot radiation — Treatment of each cycle should ideally take place on two consecutive days. Allowing for holidays, weekends, and other scheduling issues or unexpected delays, treatment may be completed within five calendar days.

SUMMARY:
The investigators propose evaluating the feasibility of using the novel cone beam computed tomography (CBCT)-guided Ethos system to deliver expedited, adaptive Quad shot radiation for the purpose of palliative radiation of patients with advanced head and neck cancers or patients with a history of any malignancy experiencing current head and neck lesions. Quad shot radiation was selected as the palliative regimen of choice given its low toxicity profile, well published efficacy in palliation, frequent usage in the US for palliation of head and neck cancers, and safety in the setting of re-irradiation. The use of the Ethos platform to perform online adaptive radiation planning and delivery remains novel and untested. The Ethos system would be used to consolidate CT simulation, replanning, and treatment for Quad shot patients receiving treatment with the benefit of reduced patient travel and a reduction in the unwanted delay between Quad shot cycles. The goal of this pilot study will be to evaluate the feasibility of the Ethos system to eliminate the need for a CT simulation for cycles 2 and 3 of Quad shot radiation.

ELIGIBILITY:
Inclusion Criteria:

* History of a head and neck malignancy or history of any malignancy experiencing current head and neck lesions suitable for radiation. Past history of radiotherapy is allowed for inclusion and brain metastases are allowed for inclusion.
* Deemed medically fit for Quad shot radiation by treating physician
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

-Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry. If pregnancy test is not clinically indicated as determined by treating physician or protocol PI, documentation of this exception is sufficient in lieu of pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the successful completion of Quad shot radiation using CBCT instead of routine CT simulation in 80% of attempted simulated patients | Completion of treatment by all patients enrolled (estimated to be 3 years and 12 weeks)

SECONDARY OUTCOMES:
Average time (days) required from initial consult to completion of radiation therapy for patient travel and visits to the department | Approximately 12 weeks
Percentage of patients from whom repeat CT simulation was eliminated | Completion of treatment by all patients enrolled (estimated to be 3 years and 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Thorstad, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide a summary of basic outcomes and clinical results within one year.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu